CLINICAL TRIAL: NCT03243370
Title: Clock'N' Test: Development and Validation (in a Control Population) of a Test Based on Time Estimations and Aiming to Evaluate Emotional Disorders
Brief Title: Clock'N' Test: Development and Validation of a Test to Evaluate Emotional Disorders
Acronym: Clock'N'test
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GROS-GIROUD-2014
Record Dates: First submitted 2017-02-02; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-01

CONDITIONS: Healthy
Keywords: Validate the Clock'nTest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study concerns the validation of a clinical test that aims to reveal "first level" emotional disorders in neurological diseases.

In order to bring to light such disorders, it is necessary to begin by establishing reference values in healthy individuals. This test is based on the priming effect and time estimations. The test procedure has two successive phases. The first phase aims to determine the judgement of time inherent to each participant and then to assess whether or not this judgement varies during the second phase with the introduction of emotional priming. First, we set out to look for and to calibrate video stimuli able to activate emotions. To this end, we used a battery of 70 sequences developed recently by Schaefer, Nils, Sanchez and Philippot. We determined their degree of physiological activation by measuring the electrodermal response at the laboratory for the exploration of the nervous system in Dijon. These measurements also allowed us to define and refine our paradigm, notably by deciding at what moment the time estimation task should be done and by eliminating the influence of attention. We decided to select only seven video sequences because we noticed a reduction in the measurement effect on time estimations due to habituation of the subject. We also conducted pre-tests in a control population made up of twenty men and women aged from 20 to 60 years.

This brought to light a warp in time estimation opposite to that we found using olfactory stimuli. This first finding suggests that there are two types of emotion, one which is anticipative and the other immediately experienced.

ELIGIBILITY:
Inclusion Criteria:

* persons who have given their consent to participate
* aged between 20 and 92 years.
* persons who understand and speak French.
* persons informed about the study

Exclusion Criteria:

* persons without national health insurance cover
* disease likely to cause emotional disorders (history of paralimbic brain tumour, MS, Parkinson, history of depression, bipolar disorder…).
* heart disease, spasmophilia.
* cognitive disorders likely to interfere with understanding the instructions.
* visual or auditory, sensory or motor disorders.
* refusal to participate in the study.

Ages: 20 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This test is based on the priming effect and time estimations. The test procedure has two successive phases. The first phase aims to determine the judgement of time inherent to each participant and then to assess whether or not this judgement varies during the second phase with the introduction of emotional priming.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Score obtained in the Clock n'test: [time estimation with priming]-[time estimation without priming]. | 1 day
  Bring to light "first-level" emotional disorders. It is based on the priming effect of time estimation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Dijon, Dijon, France

IPD SHARING:
Plan to Share IPD: No